CLINICAL TRIAL: NCT01849952
Title: Evaluating the Expression Levels of microRNA-10b in Patients With Gliomas
Status: Terminated | Type: Observational
Why Stopped: Study was administratively closed by IRB
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: D12160
Record Dates: First submitted 2013-05-06; First posted 2013-05-09 (Estimated); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Astrocytoma; Oligodendroglioma; Oligoastrocytoma; Anaplastic Astrocytoma; Anaplastic Oligodendroglioma; Anaplastic Oligoastrocytoma; Glioblastoma; Brain Tumors; Brain Cancer
Keywords: glioblastoma; miRNA; GBM; astrocytoma
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma; Glioblastoma; Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, tumor tissue, cerebrospinal fluid.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
MicroRNAs (miRNA) are molecular biomarkers that post-transcriptionally control target genes. Deregulated miRNA expression has been observed in diverse cancers. In high grade gliomas, known as glioblastomas, the investigators have identified an oncogenic miRNA, miRNA-10b (mir-10b) that is expressed at higher levels in glioblastomas than in normal brain tissue. This study tests the hypothesis that in primary glioma samples mir-10b expression patterns will serve as a prognostic and diagnostic marker. This study will also characterize the phenotypic and genotypic diversity of glioma subclasses. Furthermore, considering the critical function of anti-mir-10b in blocking established glioblastoma growth, the investigators will test in vitro the sensitivity of individual primary tumors to anti-mir-10b treatment. Tumor, blood and cerebrospinal fluid samples will be obtained from patients diagnosed with gliomas over a period of two years. These samples will be examined for mir-10b expression levels. Patient survival, as well as tumor grade and genotypic variations will be correlated to mir-10b expression levels.

ELIGIBILITY:
Inclusion/Exclusion Criteria:

* 18 years of age
* Brain tumor(s) to be resected for clinical reasons.
* Histological pathology confirmation that tumor is of glial origin, WHO Grade II, III or IV.
* Adequate tissue available for processing as determined by Pathology.
* Adequate decision making ability to review, discuss and sign a consent form to allow their tumor samples to be used for future human brain tumor biology laboratory research. Determination of capacity to consent is made by one of the co-investigators based on clinical assessment.
* Patients opting for the standard treatment regimen for their disease as well as ongoing clinical trials will be are eligible to participate in this study. Standard care for newly-diagnosed glioblastomas typically consists of surgical resection followed by radiotherapy with concomitant temozolomide, followed by adjuvant temozolomide chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seen in the clinic who are going to be treated with surgery, radiation and medical therapy for gliomas will be eligible for the study.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2013-10-09 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2025-08-25 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 24 months
  Patients will be followed for survival every 12 weeks +/- 1 week.

SECONDARY OUTCOMES:
Progression-Free Survival | 24 Months

CONTACTS AND LOCATIONS:
Overall Officials: Arti B Gaur, PhD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (4):
- United States (4):
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - University of Vermont, Burlington, Vermont

REFERENCES:
- [Background] Gaur A, Jewell DA, Liang Y, Ridzon D, Moore JH, Chen C, Ambros VR, Israel MA. Characterization of microRNA expression levels and their biological correlates in human cancer cell lines. Cancer Res. 2007 Mar 15;67(6):2456-68. doi: 10.1158/0008-5472.CAN-06-2698. PMID 17363563
- [Background] Gaur AB, Holbeck SL, Colburn NH, Israel MA. Downregulation of Pdcd4 by mir-21 facilitates glioblastoma proliferation in vivo. Neuro Oncol. 2011 Jun;13(6):580-90. doi: 10.1093/neuonc/nor033. PMID 21636706
- [Background] Sathornsumetee S, Rich JN. Designer therapies for glioblastoma multiforme. Ann N Y Acad Sci. 2008 Oct;1142:108-32. doi: 10.1196/annals.1444.009. PMID 18990124
- [Background] Lo HW. EGFR-targeted therapy in malignant glioma: novel aspects and mechanisms of drug resistance. Curr Mol Pharmacol. 2010 Jan;3(1):37-52. doi: 10.2174/1874467211003010037. PMID 20030624
- [Background] Nagarajan RP, Costello JF. Epigenetic mechanisms in glioblastoma multiforme. Semin Cancer Biol. 2009 Jun;19(3):188-97. doi: 10.1016/j.semcancer.2009.02.005. Epub 2009 Feb 20. PMID 19429483
- [Background] Quick A, Patel D, Hadziahmetovic M, Chakravarti A, Mehta M. Current therapeutic paradigms in glioblastoma. Rev Recent Clin Trials. 2010 Jan;5(1):14-27. doi: 10.2174/157488710790820544. PMID 20205684
- [Background] Stupp R, Mason WP, van den Bent MJ, Weller M, Fisher B, Taphoorn MJ, Belanger K, Brandes AA, Marosi C, Bogdahn U, Curschmann J, Janzer RC, Ludwin SK, Gorlia T, Allgeier A, Lacombe D, Cairncross JG, Eisenhauer E, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumor and Radiotherapy Groups; National Cancer Institute of Canada Clinical Trials Group. Radiotherapy plus concomitant and adjuvant temozolomide for glioblastoma. N Engl J Med. 2005 Mar 10;352(10):987-96. doi: 10.1056/NEJMoa043330. PMID 15758009
- [Background] Salcman M. Survival in glioblastoma: historical perspective. Neurosurgery. 1980 Nov;7(5):435-9. doi: 10.1227/00006123-198011000-00001. PMID 6255368
- [Background] Stewart LA. Chemotherapy in adult high-grade glioma: a systematic review and meta-analysis of individual patient data from 12 randomised trials. Lancet. 2002 Mar 23;359(9311):1011-8. doi: 10.1016/s0140-6736(02)08091-1. PMID 11937180
- [Background] Brada M, Hoang-Xuan K, Rampling R, Dietrich PY, Dirix LY, Macdonald D, Heimans JJ, Zonnenberg BA, Bravo-Marques JM, Henriksson R, Stupp R, Yue N, Bruner J, Dugan M, Rao S, Zaknoen S. Multicenter phase II trial of temozolomide in patients with glioblastoma multiforme at first relapse. Ann Oncol. 2001 Feb;12(2):259-66. doi: 10.1023/a:1008382516636. PMID 11300335
- [Background] Westphal M, Hilt DC, Bortey E, Delavault P, Olivares R, Warnke PC, Whittle IR, Jaaskelainen J, Ram Z. A phase 3 trial of local chemotherapy with biodegradable carmustine (BCNU) wafers (Gliadel wafers) in patients with primary malignant glioma. Neuro Oncol. 2003 Apr;5(2):79-88. doi: 10.1093/neuonc/5.2.79. PMID 12672279
- [Background] Holland EC, Celestino J, Dai C, Schaefer L, Sawaya RE, Fuller GN. Combined activation of Ras and Akt in neural progenitors induces glioblastoma formation in mice. Nat Genet. 2000 May;25(1):55-7. doi: 10.1038/75596. PMID 10802656
- [Background] Sonoda Y, Ozawa T, Hirose Y, Aldape KD, McMahon M, Berger MS, Pieper RO. Formation of intracranial tumors by genetically modified human astrocytes defines four pathways critical in the development of human anaplastic astrocytoma. Cancer Res. 2001 Jul 1;61(13):4956-60. PMID 11431323
- [Background] Furnari FB, Fenton T, Bachoo RM, Mukasa A, Stommel JM, Stegh A, Hahn WC, Ligon KL, Louis DN, Brennan C, Chin L, DePinho RA, Cavenee WK. Malignant astrocytic glioma: genetics, biology, and paths to treatment. Genes Dev. 2007 Nov 1;21(21):2683-710. doi: 10.1101/gad.1596707. PMID 17974913
- [Background] Dell'Albani P. Stem cell markers in gliomas. Neurochem Res. 2008 Dec;33(12):2407-15. doi: 10.1007/s11064-008-9723-8. Epub 2008 May 21. PMID 18493853
- [Background] Standart N, Jackson RJ. MicroRNAs repress translation of m7Gppp-capped target mRNAs in vitro by inhibiting initiation and promoting deadenylation. Genes Dev. 2007 Aug 15;21(16):1975-82. doi: 10.1101/gad.1591507. No abstract available. PMID 17699746
- [Background] de Moor CH, Meijer H, Lissenden S. Mechanisms of translational control by the 3' UTR in development and differentiation. Semin Cell Dev Biol. 2005 Feb;16(1):49-58. doi: 10.1016/j.semcdb.2004.11.007. Epub 2005 Jan 12. PMID 15659339
- [Background] Zhang B, Wang Q, Pan X. MicroRNAs and their regulatory roles in animals and plants. J Cell Physiol. 2007 Feb;210(2):279-89. doi: 10.1002/jcp.20869. PMID 17096367
- [Background] Miska EA. How microRNAs control cell division, differentiation and death. Curr Opin Genet Dev. 2005 Oct;15(5):563-8. doi: 10.1016/j.gde.2005.08.005. PMID 16099643
- [Background] Sevignani C, Calin GA, Siracusa LD, Croce CM. Mammalian microRNAs: a small world for fine-tuning gene expression. Mamm Genome. 2006 Mar;17(3):189-202. doi: 10.1007/s00335-005-0066-3. Epub 2006 Mar 3. PMID 16518686
- [Background] Louis DN, Ohgaki H, Wiestler OD, Cavenee WK, Burger PC, Jouvet A, Scheithauer BW, Kleihues P. The 2007 WHO classification of tumours of the central nervous system. Acta Neuropathol. 2007 Aug;114(2):97-109. doi: 10.1007/s00401-007-0243-4. Epub 2007 Jul 6. PMID 17618441
- See also: Norris Cotton Cancer Center Clinical Trial Page — https://cancer.dartmouth.edu/patients-families/find-clinical-trial/trial/D12160